CLINICAL TRIAL: NCT04024943
Title: Personalized Therapy Study - Attain Stability Quad Post-Approval Study
Acronym: ASQ
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Attain Stability Quad PAS
Record Dates: First submitted 2019-06-24; First posted 2019-07-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Quadripolar LV Lead — The Attain Stability Quad MRI SureScan LV Lead (Model 4798) is an active fixation quadripolar LV lead based on the Attain Performa lead family models (4298, 4398, and 4598). The lead incorporates an active fixation helix similar to the OUS commercialized Attain Stability bipolar LV lead (Model 20066/4796) which is designed to allow an implanter more options in lead location.
  Other Names: Medtronic CRT-P; Medtronic CRT-D

SUMMARY:
The purpose of this Post-Approval Study (PAS) is to evaluate the long-term performance of the Model 4798 Left Ventricular (LV) lead in a real-world patient population. Patients will be followed for the duration of the PAS. This study is required by FDA as a condition of approval of the Model 4798 LV lead and is integrated within the Product Surveillance Registry (PSR).

DETAILED DESCRIPTION:
The Attain Stability Quad (ASQ) PAS is a multi-center, single arm, prospective observational study. However, in the US, retrospective enrollments from participants in the IDE study (IDE #G170020) are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive or be treated with a Model 4798 lead and a Medtronic CRT device
* Patient within 30 days of therapy received at the time of their initial PSR platform enrollment

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients that are or will be implanted with a Model 4798 lead and a Medtronic CRT device.
Sampling Method: Non-Probability Sample
Enrollment: 1092 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients without a lead- related event at 5 years post-implant | 5 years
  To demonstrate that the complication-free probability is greater than 92.5% at five years post-implant for Attain Stability Quad LV leads.

SECONDARY OUTCOMES:
Number of lead-related adverse device effects | 5 years
  The secondary objectives are descriptive in nature and are intended to gain additional information about the safety and performance of the Product:
  • To summarize all Attain Stability Quad lead-related ADEs
Number of explanted leads that have been returned | 5 years
  The secondary objectives are descriptive in nature and are intended to gain additional information about the safety and performance of the Product:
  • To summarize analysis results from explanted and returned Attain Stability Quad leads

CONTACTS AND LOCATIONS:
Locations (115):
- United States (72):
  - Alaska Heart, Anchorage, Alaska
  - Southwest EP, Chandler, Arizona
  - Cardiology Associates of Northeast Arkansas, Jonesboro, Arkansas
  - Saint Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - Chula Vista Cardiac Center, Chula Vista, California
  - San Diego Arrhythmia Associates, San Diego, California
  - COR Healthcare, Torrance, California
  - Cardiovascular Consultants Medical Group (Van Nuys), Van Nuys, California
  - Cardiology Associates Medical Group, Ventura, California
  - Colorado Springs Cardiology, Colorado Springs, Colorado
  - Denver Heart, Denver, Colorado
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Heart Rhythm Solutions, Hollywood, Florida
  - Baptist Health, Jacksonville, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Heart & Vascular Institute of Florida, Safety Harbor, Florida
  - Heart Rhythm Consultants P.A. (Sarasota Memorial Research), Sarasota, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Deaconess Specialty Physicians, Evansville, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Saint Elizabeth Healthcare, Edgewood, Kentucky
  - Norton Heart Specialists, Louisville, Kentucky
  - Our Lady of the Lake Office of Research, Baton Rouge, Louisiana
  - MedStar Health Research Institute, Baltimore, Maryland
  - Tidal Health Peninsula Regional, Salisbury, Maryland
  - Associates in Cardiology PA, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital (Boston, MA), Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - UP Health System - Marquette, Marquette, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - North Memorial Heart and Vascular Institute, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - University Hospital of Missouri, Columbia, Missouri
  - Saint Lukes Health System, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Nebraska Medicine, Omaha, Nebraska
  - Monmouth Cardiology Associates, Ocean City, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - South Shore University Hospital, Bay Shore, New York
  - Huntington Hospital, Huntington, New York
  - North Shore University Hospital, Manhasset, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - New York-Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Staten Island University Hospital, Staten Island, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Summa Center for Clinical Trials-Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - The Christ Hospital Health Network, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Heart and Vascular Institute at UPMC Hamot, Erie, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Heart Center of North Texas, Fort Worth, Texas
  - Consultants in Cardiology, Fort Worth, Texas
  - EP Heart, The Woodlands, Texas
  - Kootenai Heart Clinics Northwest, Spokane, Washington
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- France (13):
  - Clinique Rhône Durance, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHRU Brest - Hôpital de la Cavale Blanche, Brest
  - Générale de Santé - Hôpital Privé Saint Martin, Caen
  - CHU de Caen - Hôpital Côte de Nacre - Centre Esquirol, Caen
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU de Dijon - Hospital Le Bocage, Dijon
  - CHRU La Rochelle, La Rochelle
  - Hopital prive Clairval - Ramsay Sante, Marseille
  - Nouvelles Cliniques Nantaises, Nantes
  - Centre hospitalier de la région d'Annecy, Pringy
  - Centre Hospitalier Universitaire Saint Étienne - Hôpital Nord, Saint-Priest-en-Jarez
  - Capio - Clinique du Tonkin, Villeurbanne
- Greece (2):
  - Hygeia Hospital, Athens
  - Athens Medical Center, Marousi
- Italy (6):
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - Azienda Sanitaria Provinciale di Cosenza "Ospedale di Castrovillari", Castrovillari
  - Ospedale "Vito Fazzi" Lecce, Lecce
  - Azienda Ospedaliera Ospedale Niguarda Ca Granda, Milan
  - Presidio Ospedaliero Centrale - SS. Annunziata, Taranto
  - Azienda ospedaleria Santa Maria della Misericordia di Udine, Udine
- Portugal (4):
  - Hospital da Senhora da Oliveira - Guimarães, Guimarães
  - Hospital de Santa Maria-Centro Hospitalar Lisboa Norte, EPE, Lisbon
  - Centro Hospitalar Universitário de São João, Porto
  - Hospital Distrital de Santarém, Santarém
- Národný ústav srdcových a cievnych chorôb, a.s. (NUSCH, a.s.), Bratislava, Slovakia
- Spain (8):
  - Hospital Universitario da Coruna, A Coruña
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Switzerland (2):
  - Hôpitaux Universitaires de Genève, Geneva
  - Cardiopark Zurich, Zurich
- United Kingdom (7):
  - University Hospitals of Birmingham NHS Foundation Trust - Queen Elizabeth Hospital, Birmingham
  - Blackpool, Fylde and Wyre Hospitals NHS Foundation Trust - Blackpool Victoria Hospital, Blackpool
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London
  - Central Manchester University Hospitals NHS - Manchester Royal Infirmary, Manchester
  - The James Cook University Hospital - South Tees Hospitals NHS, Middlesbrough
  - Sheffield Vascular Institute, Sheffield Teaching Hospitals NHS - Northern General, Sheffield

IPD SHARING:
Plan to Share IPD: No